CLINICAL TRIAL: NCT00912093
Title: A Phase III Randomized, Double-Blind,Placebo-Controlled, Multicenter Study of Icatibant for Subcutaneous Injection in Patients With Acute Attacks of Hereditary Angioedema (HAE)
Brief Title: A Study of Icatibant in Patients With Acute Attacks of Hereditary Angioedema (FAST-3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HGT-FIR-054; 2009-015606-19 (EudraCT Number)
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Results first posted 2014-08-06 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Hereditary Angioedema
Keywords: HAE; Type I HAE; Type II HAE
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — icatibant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Single subcutaneous injection of matching placebo
  Interventions: Drug: Placebo
- Icatibant (Experimental): Single subcutaneous injection of icatibant, 30 mg
  Interventions: Drug: Icatibant

INTERVENTIONS:
Drug: Icatibant — Single subcutaneous injection of icatibant, 30 mg
  Other Names: Firazyr
  Arms: Icatibant
Drug: Placebo — Single subcutaneous injection of matching placebo
  Arms: Placebo

SUMMARY:
This study is being conducted to evaluate the efficacy and safety of icatibant compared to placebo in patients experiencing acute attacks of hereditary angioedema (HAE).

DETAILED DESCRIPTION:
This Phase III study consisted of two parts: A controlled phase and an open label extension (OLE) phase.

The controlled phase describes the double blind part of the study and was intended to evaluate the efficacy and safety of icatibant compared with placebo for the first treated cutaneous and/or abdominal attack.

Patients with moderate to severe abdominal or cutaneous attacks were randomized to receive a single, blinded, subcutaneous injection of icatibant (30 mg) or placebo. After a protocol amendment, patients with mild to moderate laryngeal HAE attacks were also randomized to receive a single, blinded subcutaneous injection of icatibant (30 mg) or placebo in order to obtain blinded, controlled efficacy and safety data for this subset of subjects. Patients experiencing severe laryngeal attacks (post-amendment) or mild to severe laryngeal attacks (pre-amendment) were to receive open-label icatibant.

After treatment of the first attack in the controlled phase, patients were eligible to enter the OLE phase. In the OLE phase, patients who experienced angioedema attacks severe enough to warrant treatment were to be treated with s.c. icatibant as appropriate until the study was discontinued or the product was commercially available.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet the following criteria to be enrolled in this study.

1. The patient is ≥18 years old at the time of informed consent.
2. The patient has a documented diagnosis of HAE type I or II. The diagnosis will be confirmed either by documented decreased C4 levels and/or immunogenic or functional C1-INH deficiency results (<50% of normal levels) consistent with HAE types I and II or by medical history.
3. The current HAE attack must be in the cutaneous, abdominal and/or laryngeal (inclusive of laryngeal and pharyngeal) areas.
4. Cutaneous or abdominal HAE attacks must be moderate to very severe as determined by investigator global assessment at pre-treatment assessments
5. The patient must report at least 1 VAS score ≥ 30mm
6. The patient commences treatment within 6 hours of the attack becoming at least mild (laryngeal) or moderate (non-laryngeal) in severity, but not more than 12 hours after the onset of the attack.
7. Women of childbearing potential must have a negative urine pregnancy test and must use appropriate methods to prevent pregnancy during their participation in the study.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study.

1. The patient has a diagnosis of angioedema other than HAE type I or II.
2. The patient has received previous treatment with icatibant.
3. The patient has participated in a clinical trial and has received treatment with another investigational medicinal product within the past 30 days.
4. The patient has received treatment with any pain medication since the onset of the current angioedema attack.
5. The patient has received replacement therapy (fresh frozen plasma [FFP], C1-INH products) less than 5 days (120 hours) from the onset of the current angioedema attack.
6. The patient is receiving treatment with angiotensin converting enzyme (ACE) inhibitors.
7. Evidence of coronary artery disease based on medical history or screening examination in particular unstable angina pectoris or severe coronary heart disease;
8. The patient has a serious concomitant illness or condition that, in the opinion of the Investigator, would be a contraindication for participation in the trial.
9. The patient is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2009-07-16 (Actual); Primary Completion 2010-10-01 (Actual); Study Completion 2010-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (64):
- United States (39):
  - Primary Care Associates of Alabaster, Alabaster, Alabama
  - UAB Lung Health Center, Birmingham, Alabama
  - Medical Research of AZ A Division of Allergy & Immunology Assoc, Scottsdale, Arizona
  - Little Rock Allergy & Asthma Clinic, PA, Little Rock, Arkansas
  - Allergy and Asthma Insititute of the Valley, Granada Hills, California
  - University of California San Diego, La Jolla, California
  - UCLA - Clinical Immunology & Allergy, Los Angeles, California
  - Speciality Medical Clinic & Research Center, Stanford, California
  - Standford University, Stanford, California
  - Asthma & Allergy Associates, PC, Colorado Springs, Colorado
  - Medical Associates of Brevard, Melbourne, Florida
  - University of South Florida Division of Allergy and Immunology, Tampa, Florida
  - Family Allergy and Asthma Center, PC, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Research Institute of Deaconess Clinic, Evansville, Indiana
  - University of Iowa Asthma Center/ Hospitals & Clinics, Iowa City, Iowa
  - LSUHSC Allergy & Immunology, Shreveport, Louisiana
  - Institute for Asthman & Allergy, P.C., Chevy Chase, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Asthma Center, St Louis, Missouri
  - University of Reno Nevada School of Medicine, Reno, Nevada
  - STARx Research Center, LLC, Edison, New Jersey
  - Winthrop University Hospital Clinical Trials Center, Mineola, New York
  - Mount Sinai School of Medicine, New York, New York
  - Montefiore Medical Center/Albert Einstein College of Medicine, The Bronx, New York
  - Allergy Partners of Western North Carolina, Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Division of Immunology/Allergy, Cincinnati, Ohio
  - Optimed Research, LTD, Columbus, Ohio
  - Tulsa Allergy Clinic, Tulsa, Oklahoma
  - Baker Allergy, Asthma & Dermatology Research Center LLC, Lake Oswego, Oregon
  - Valley Clinical Research Center, Bethlehem, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Pittsburgh (of UMPC), Pittsburgh, Pennsylvania
  - AARA Research Center, Dallas, Texas
  - University of Texas Medical Branch (UTMB), Galveston, Texas
  - Texas A&M Health Science Center College of Medicine, Houston, Texas
  - Allergy and Asthma Research Center, P.A., San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
- Australia (4):
  - Canberra Hospital Department of Immunology, Garran, Australian Capital Territory
  - Dept of Medicine Immunology & Allergy Campbelltown Hospital, Campbelltown, New South Wales
  - Royal Melbourne Hospital Department of Immunology, Parkville, Victoria
  - Royal Adelaide Hospital, Adelaide
- Canada (3):
  - NACTRC, Edmonton, Alberta
  - Allergy & Asthma Research Centre, Ottawa, Ontario
  - Centre de recherché Appliquée en allergie de Québec, Québec, Quebec
- 3rd Department of Internal Medicine Semmelweis University, Budapest, Hungary
- Israel (3):
  - Bnai-Zion Medical Center Division of Immunology & Allergy, Haifa
  - Tel Aviv Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Spitalul Clinic Judetean Mures Sectia Medicina Interna, Târgu Mureş, Transylvania, Romania
- Russia (7):
  - Medical Academy of Postgraduate Education, Saint Petersburg, Sankt-Peterburg
  - Autonomous Non Commercial Organization, Saint Petersburg, Sankt-Peterburg
  - State Healthcare Institution of City of Moscow, Moscow
  - State Enterprise State Scientific Centre, Moscow
  - State Educational Institution of Additional Profess. Edu. Moscow, Moscow
  - Municipal Medical & Preventive Treatment Institution, Smolensk
  - Regional Clinical Center of Specialized Medical Treatment, Vladivostok
- Allergy Diagnostic and Clinical Research Unit (ADCRU), Cape Town, Mowbray, South Africa
- Ukraine (5):
  - Ivano-Frankivsk national Medical University, Ivano-Frankivsk
  - National Medical Academy for Postgraduate Education, Kyiv
  - Institute of Otolaryngology, Kyiv
  - Ukranian Medical Stomatological Academy Dept of Int Diseases, Poltava
  - Vinnitsa Medical Academy Chair of Internal Disease, Vinnitsa

REFERENCES:
- [Derived] Lumry WR, Farkas H, Moldovan D, Toubi E, Baptista J, Craig T, Riedl M. Icatibant for Multiple Hereditary Angioedema Attacks across the Controlled and Open-Label Extension Phases of FAST-3. Int Arch Allergy Immunol. 2015;168(1):44-55. doi: 10.1159/000441060. Epub 2015 Nov 11. PMID 26556097
- [Derived] Maurer M, Longhurst HJ, Fabien V, Li HH, Lumry WR. Treatment of hereditary angioedema with icatibant: efficacy in clinical trials versus effectiveness in the real-world setting. Allergy Asthma Proc. 2014 Sep-Oct;35(5):377-81. doi: 10.2500/aap.2014.35.3780. Epub 2014 Aug 6. PMID 25198193
- [Derived] Bas M. Clinical efficacy of icatibant in the treatment of acute hereditary angioedema during the FAST-3 trial. Expert Rev Clin Immunol. 2012 Nov;8(8):707-17. doi: 10.1586/eci.12.67. PMID 23167682
- [Derived] Lumry WR, Li HH, Levy RJ, Potter PC, Farkas H, Moldovan D, Riedl M, Li H, Craig T, Bloom BJ, Reshef A. Randomized placebo-controlled trial of the bradykinin B(2) receptor antagonist icatibant for the treatment of acute attacks of hereditary angioedema: the FAST-3 trial. Ann Allergy Asthma Immunol. 2011 Dec;107(6):529-37. doi: 10.1016/j.anai.2011.08.015. Epub 2011 Oct 5. PMID 22123383

RESULTS

PARTICIPANT FLOW:
Groups:
- Randomized-Icatibant (Blinded Treatment)-Non-laryngeal: Subjects with moderate to severe cutaneous or abdominal attacks of HAE randomized to receive a single subcutaneous injection of icatibant, 30 mg in the controlled phase
- Randomized-Placebo (Blinded Treatment)-Non-laryngeal: Subjects with moderate to severe cutaneous or abdominal attacks of HAE randomized to receive a single subcutaneous injection of matching placebo in the controlled phase
- Randomized-Icatibant (Blinded Treatment)-Laryngeal: Subjects with mild to moderate laryngeal attacks of HAE randomized to receive a single subcutaneous injection of icatibant, 30 mg in the controlled phase
- Randomized-Placebo (Blinded Treatment)-Laryngeal: Subjects with mild to moderate laryngeal attacks of HAE randomized to receive a single subcutaneous injection of matching placebo in the controlled phase
- Open-Label Icatibant-Severe Laryngeal: Subjects with severe (post-amendment) or mild to severe (pre-amendment) laryngeal attacks of HAE treated with subcutaneous injection of icatibant, 30 mg in the controlled phase
Period: The Controlled Phase
Arm/Group | Randomized-Icatibant (Blinded Treatment)-Non-laryngeal | Randomized-Placebo (Blinded Treatment)-Non-laryngeal | Randomized-Icatibant (Blinded Treatment)-Laryngeal | Randomized-Placebo (Blinded Treatment)-Laryngeal | Open-Label Icatibant-Severe Laryngeal
Started | 43 | 45 | 3 | 2 | 5
Completed | 43 | 43 | 3 | 2 | 4
Not Completed | 0 | 2 | 0 | 0 | 1
Not completed — Death | 0 | 1 | 0 | 0 | 0
Not completed — Medical Condition | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Period: The Open Label Extension (OLE) Phase
Arm/Group | Randomized-Icatibant (Blinded Treatment)-Non-laryngeal | Randomized-Placebo (Blinded Treatment)-Non-laryngeal | Randomized-Icatibant (Blinded Treatment)-Laryngeal | Randomized-Placebo (Blinded Treatment)-Laryngeal | Open-Label Icatibant-Severe Laryngeal
Started | 38 | 35 | 3 | 2 | 4
Completed | 38 | 35 | 3 | 2 | 4
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Randomized-Icatibant (Blinded Treatment)--Non-laryngeal: Subjects with moderate to severe cutaneous or abdominal attacks of HAE randomized to receive a single subcutaneous injection of icatibant 30 mg in the controlled phase
- Randomized-Icatibant (Blinded Treatment)--Laryngeal: Subjects with mild to moderate laryngeal attacks of HAE randomized to receive a single subcutaneous injection of icatibant 30 mg in the controlled phase
- Open-Label Icatibant-Severe Laryngeal: Subjects with severe (post-amendment) or mild to severe (pre-amendment) laryngeal attacks of HAE treated with subcutaneous injection of icatibant 30 mg in the controlled phase
- Total: Total of all reporting groups
Arm/Group | Randomized-Icatibant (Blinded Treatment)--Non-laryngeal | Randomized-Placebo (Blinded Treatment)-Non-laryngeal | Randomized-Icatibant (Blinded Treatment)--Laryngeal | Randomized-Placebo (Blinded Treatment)-Laryngeal | Open-Label Icatibant-Severe Laryngeal | Total
Number analyzed (Participants) | 43 | 45 | 3 | 2 | 5 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (13.69) | 36.6 (11.18) | 40.3 (6.66) | 50.0 (22.63) | 41.6 (11.78) | 37.0 (12.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 29 | 2 | 1 | 2 | 61
  Male | 16 | 16 | 1 | 1 | 3 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific | 0 | 0 | 0 | 0 | 0 | 0
  White | 38 | 40 | 3 | 2 | 4 | 87
  Other | 2 | 5 | 0 | 0 | 1 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 32 | 2 | 2 | 3 | 65
  Hungary | 3 | 1 | 0 | 0 | 0 | 4
  Canada | 1 | 0 | 0 | 0 | 0 | 1
  Ukraine | 0 | 1 | 0 | 0 | 0 | 1
  Romania | 3 | 1 | 1 | 0 | 0 | 5
  Australia | 2 | 3 | 0 | 0 | 0 | 5
  Russian Federation | 2 | 1 | 0 | 0 | 0 | 3
  South Africa | 2 | 1 | 0 | 0 | 1 | 4
  Israel | 4 | 5 | 0 | 0 | 1 | 10
Weight (kg) [Count of Participants; unit: Participants]
  <= 50 kg | 4 | 2 | 0 | 0 | 0 | 6
  >50-75 kg | 16 | 20 | 1 | 2 | 0 | 39
  >75-100 kg | 14 | 13 | 1 | 0 | 3 | 31
  >100 kg | 9 | 10 | 1 | 0 | 2 | 22

OUTCOME MEASURES:

1. Primary Outcome: Time to Onset of Symptom Relief for an Acute Attack, as Assessed by the Patient
Description: Time to onset of symptom relief was calculated from study drug administration to onset of symptom relief, where onset of symptom relief was defined as the earliest of 3 consecutive measurements in which there was a 50% reduction from pretreatment in composite VAS score. Composite VAS score comprised 3 symptoms, including skin swelling, skin pain, and abdominal pain, for cutaneous and abdominal attacks and 5 symptoms, including skin swelling, skin pain, abdominal pain, difficulty swallowing, and voice change, for laryngeal attacks. Subjects who did not achieve symptom relief within the observation period were censored at the last observation time.
Time Frame: Up to 120 hours post-dose
Population: Non-laryngeal Intent-to-Treat (nl-ITT) population included all subjects with non-laryngeal attacks of HAE randomized to treatment. Subjects were analyzed according to the randomized treatment regardless of the treatment actually received. This was the primary analysis population for efficacy.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Randomized-Icatibant (Blinded Treatment)--Non-laryngeal | Randomized-Placebo (Blinded Treatment)-Non-laryngeal
Number analyzed (Participants) | 43 | 45
Hours | 2.0 [1.5 to 3.0] | 19.8 [6.1 to 26.3]
Statistical Analysis 1: Comparison: Randomized-Icatibant (Blinded Treatment)--Non-laryngeal vs Randomized-Placebo (Blinded Treatment)-Non-laryngeal; Test type: Superiority or Other; p < 0.001, Peto-Peto Wilcoxon

2. Secondary Outcome: Time to Onset of Primary Symptom Relief
Description: Time to primary symptom relief was calculated from the time of study drug administration to the onset of primary symptom relief, where onset of primary symptom relief was determined using the subject-assessed VAS score for a single primary symptom (determined by edema location) and defined as the earliest of 3 consecutive non-missing measurements in which a pre-specified reduction from the pretreatment value was met. Subjects who did not achieve primary symptom relief within the observation period were censored at the last observation time.
Time Frame: Up to 120 hours post-dose
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Randomized-Icatibant (Blinded Treatment)--Non-laryngeal | Randomized-Placebo (Blinded Treatment)-Non-laryngeal
Number analyzed (Participants) | 43 | 45
Hours | 1.5 [1.0 to 2.0] | 18.5 [3.6 to 23.9]
Statistical Analysis 1: Comparison: Randomized-Icatibant (Blinded Treatment)--Non-laryngeal vs Randomized-Placebo (Blinded Treatment)-Non-laryngeal; Test type: Superiority or Other; p < 0.001, Peto-Peto Wilcoxon

3. Secondary Outcome: Time to Almost Complete Symptom Relief
Description: Time to almost complete symptom relief was calculated from the time of study drug administration to almost complete symptom relief, where almost complete symptom relief was defined as the earliest of 3 consecutive non-missing measurements in which all VAS scores <10 mm. Subjects who did not achieve almost complete symptom relief within the observation period were censored at the last observation time.
Time Frame: Up to 120 Hours post treatment
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Randomized-Icatibant (Blinded Treatment)--Non-laryngeal | Randomized-Placebo (Blinded Treatment)-Non-laryngeal
Number analyzed (Participants) | 43 | 45
Hours | 8.0 [5.0 to 42.5] | 36.0 [29.0 to 50.9]
Statistical Analysis 1: Comparison: Randomized-Icatibant (Blinded Treatment)--Non-laryngeal vs Randomized-Placebo (Blinded Treatment)-Non-laryngeal; Test type: Superiority or Other; p = 0.012, Peto Peto Wilcoxon

4. Secondary Outcome: Time to Subject-Assessed Initial Symptom Improvement
Description: Time to initial symptom improvement was calculated from the time of study drug administration to initial symptom improvement as determined by the subject as the time they felt symptoms were starting to improve. Subjects who did not achieve initial symptom improvement within the observation period were censored at the last observation time.
Time Frame: Up to 120 hours post-dose
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Randomized-Icatibant (Blinded Treatment)--Non-laryngeal | Randomized-Placebo (Blinded Treatment)-Non-laryngeal
Number analyzed (Participants) | 43 | 45
Hours | 0.8 [0.5 to 1.0] | 3.5 [1.9 to 5.4]
Statistical Analysis 1: Comparison: Randomized-Icatibant (Blinded Treatment)--Non-laryngeal vs Randomized-Placebo (Blinded Treatment)-Non-laryngeal; Test type: Superiority or Other; p < 0.001, Peto-Peto Wilcoxon

5. Secondary Outcome: Time to Investigator-Assessed Initial Symptom Improvement
Description: Time to initial symptom improvement was calculated from the time of study drug administration to initial symptom improvement as determined by the investigator as the time they felt symptoms were starting to improve. Subjects who did not achieve initial symptom improvement within the observation period were censored at the last observation time.
Time Frame: Up to 120 hours post-dose
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Randomized-Icatibant (Blinded Treatment)--Non-laryngeal | Randomized-Placebo (Blinded Treatment)-Non-laryngeal
Number analyzed (Participants) | 43 | 45
Hours | 0.8 [0.6 to 1.3] | 3.4 [2.6 to 6.0]
Statistical Analysis 1: Comparison: Randomized-Icatibant (Blinded Treatment)--Non-laryngeal vs Randomized-Placebo (Blinded Treatment)-Non-laryngeal; Test type: Superiority or Other; p < 0.001, Peto-Peto Wilcoxon

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events occurring within 16 days of study drug administration are included in the analysis
Description: Subjects were analyzed according to the treatment actual received
Groups:
- Controlled Phase - Icatibant (Randomized): Subjects who were randomized to treatment and received a single subcutaneous injection of icatibant 30 mg in the controlled phase
- Controlled Phase -Placebo (Randomized): Subjects who were randomized to treatment and received a single subcutaneous injection of matching placebo in the controlled phase
- Controlled Phase - Icatibant (Open Label): Subjects who were not randomized and received a single subcutaneous injection of icatibant 30 mg in the controlled phase
- Open Label Extension - Icatibant (Open Label): Subjects who treated with icatibant 30 mg in the open label extension phase
Arm/Group | Controlled Phase - Icatibant (Randomized) | Controlled Phase -Placebo (Randomized) | Controlled Phase - Icatibant (Open Label) | Open Label Extension - Icatibant (Open Label)
Serious Adverse Events (participants affected / at risk) | 0/46 | 5/46 | 0/6 | 7/82
Other Adverse Events (participants affected / at risk) | 8/46 | 12/46 | 0/6 | 23/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Controlled Phase - Icatibant (Randomized) (N=46) | Controlled Phase -Placebo (Randomized) (N=46) | Controlled Phase - Icatibant (Open Label) (N=6) | Open Label Extension - Icatibant (Open Label) (N=82)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hereditary angioedema (Congenital, familial and genetic disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tracheostomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Controlled Phase - Icatibant (Randomized) (N=46) | Controlled Phase -Placebo (Randomized) (N=46) | Controlled Phase - Icatibant (Open Label) (N=6) | Open Label Extension - Icatibant (Open Label) (N=82)
Hereditary angioedema (Congenital, familial and genetic disorders) | 5 (5) | 9 (9) | 0 (0) | 11 (17)
Headache (Nervous system disorders) | 3 (4) | 3 (3) | 0 (0) | 9 (12)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Shire's agreements with investigators vary. All agreements provide Shire the right to embargo communications regarding trial results prior to public release for a period ≤180 days from the time submitted to Shire for review. Shire does not prohibit publication, but can require the removal of confidential information (excluding trial results) and can request postponement of a single-center publication until after disclosure of the trial's multi-center publication.